CLINICAL TRIAL: NCT05443152
Title: The Effect of Self-made Fetal Movement and Position Tracking During Pregnancy on Maternal Attachment in the Postpartum Period
Brief Title: The Effect of Self-made Fetal Movement and Position Tracking During Pregnancy on Maternal Attachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AYSUN BADEM (Other)
Responsible Party: Sponsor-Investigator, AYSUN BADEM, Assistant Professor, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Maternal attachment
Record Dates: First submitted 2022-06-27; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-07

CONDITIONS: Maternal Behavior; Attachment
Keywords: Attachment; Pregnancy; Maternal attachment
MeSH Terms: interventions — Fetal Movement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arms (Experimental): Prenatal attachment scale answered. In the first stage, pregnant women were trained to implement fetal movement count and position tracking. The training was provided face to face and lasted 30-45 minutes. How to determine the position of the fetus and I. and II. Leopold maneuvers are also taught. In the second stage, the pregnant women were interviewed twice a week by telephone.Thus, it was provided that pregnant women had fetal tracked at least once a day, at any time of the day, when the fetus was awake and most active, in a suitable position and a comfortable environment, for at least 15-20 minutes continuously for four weeks. Pregnant women phoned the researcher when they wanted. At the same time, the participants continued to their routine prenatal care. The mother attachment scale was answered at least 1 month after the birth of the women.
  Interventions: Behavioral: Fetal movement and position tracking training
- No İntervention Arms (No Intervention): Prenatal attachment scale answered. The pregnant women continued to their routine prenatal care. No intervention was applied to the pregnant women in addition to their routine prenatal care.The pregnant women were called about whether continuing their routine care or having any problems during the research. The mother attachment scale was answered at least 1 month after the birth of the women.

INTERVENTIONS:
Behavioral: Fetal movement and position tracking training — In the first stage, pregnant women were trained to implement fetal movement count and position tracking. The training was provided face to face and lasted 30-45 minutes. How to determine the position of the fetus and I. and II. Leopold maneuvers are also taught. In the second stage, the pregnant women were interviewed twice a week by telephone.Thus, it was provided that pregnant women had fetal tracked at least once a day, at any time of the day, when the fetus was awake and most active, in a suitable position and a comfortable environment, for at least 15-20 minutes continuously for four weeks. Pregnant women phoned the researcher when they wanted. At the same time, the participants continued to their routine prenatal care.
  Arms: Experimental Arms

SUMMARY:
This study was conducted to determine the effect of self-made fetal movement counting and fetal position tracking on maternal attachment in prenatal period.

DETAILED DESCRIPTION:
The first attachment between mother and baby begins in the prenatal period. It is expected to increase as pregnancy progresses.The more the mother tries to communicate and interact with her baby, the stronger her attachment to her baby. The baby can be accepted by the mother as an individual, and the attachment between the mother and baby can increase.The early development of safe and positive attachment composes the basis of healthy development. In the later years of childhood, safe attachment is effective on healthy processes, such as being more positive, establishing close, constructive and respectful relationships, and a high sense of trust, while unsafe attachment is associated with emotional, social, physical and mental psychopathologies. The mother's touching her baby over her abdomen, trying to guess the parts of the baby, following baby movements, communicating with the baby by focusing and spending private time with the baby increase the physical and psychological contact with the baby. Fetal movement counting is defined as tracking uninterrupted fetal movements for at least 15-20 minutes by lying on the left side in a calm environment at any time during the day when this baby is awake. Fetal position tracking is described as trying to guess the parts of the baby by placing the mother's hand on the abdomen. In the literature, it is stated that prenatal attachment affects postpartum maternal attachment, contributes positively to infant care and provides rapid adaptation to motherhood. In addition, secure/insecure attachment styles are thought to be associated with postpartum depression. It is stated that the babies of mothers with strong prenatal attachment show healthier growth and development and even affect their personality positively in adulthood. In the literature, it is stated that the prenatal period can be an indicator of mother-infant interaction in the postpartum period.This study was carried out as a continuation of the previous study, NCT05313113 Clinical ID, to determine maternal attachment in the postpartum period of pregnant women whose fetal movement and position were followed.

ELIGIBILITY:
Inclusion Criteria:

* literate
* between the ages of 19-35
* Effective communication
* first pregnancy
* having a single fetus
* Pregnancy week between 24 and 28. between the ages of 19-35
* Effective communication
* first pregnancy
* having a single fetus
* Pregnancy week between 24 and 28.

Exclusion Criteria:

* Pregnancy using assisted reproductive techniques
* Having a risky pregnancy (preeclampsia, placenta previa, gestational diabetes etc.)
* Pregnant women with a chronic disease (heart, systemic, circulatory disorder, psychiatric, etc.) were not included in the study.

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — focused on pregnancy women
Enrollment: 85 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Prenatal attachment inventory (PAI) | between 24-28 gestational weeks and after 30 days
  The mean prenatal attachment level (mean±SD) The mean prenatal attachment was assessed using ''Prenatal attachment inventory''. The inventory consists of 21 Likert-type items. Each item is scored between 1 and 4. Therefore, the minimum score of the inventory is 21, while the maximum score of the inventory is 84. The pregnant between 24-28 gestational weeks were filled with face-to-face interviews at the first interview and 30 days after the training. [Time Frame: between 24-28 gestational weeks and after 30 days]

SECONDARY OUTCOMES:
Maternal attachment inventory (MAI) | 1-6 months after birth
  The mean maternal attachment was assessed using ''Maternal attachment inventory (MAI)''. The inventory consists of 26 Likert-type items. Each item is scored between 1 and 4. Therefore, the minimum score of the inventory is 26, while the maximum score of the inventory is 104. A high score indicates high maternal attachment. The scale can be applied between 1 month and 24 months postpartum. The scale was answered via telephone.

CONTACTS AND LOCATIONS:
Overall Officials: Aysun BADEM, asst. prof., Principal Investigator — ERCİYES UNIVERSİTY
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)